CLINICAL TRIAL: NCT00550381
Title: Ascending Single-Dose Study of the Safety, Tolerability, and Pharmacokinetics of HKI-357 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating the Safety, Tolerability, and Pharmacokinetics (PK) of HKI-357 Administered Orally to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3235A1-1000
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 1 (Placebo Comparator): 10mg
  Interventions: Drug: HKI-357
- 2 (Placebo Comparator): 20mg
  Interventions: Drug: HKI-357
- 3 (Placebo Comparator): 40mg
  Interventions: Drug: HKI-357
- 4 (Placebo Comparator): 80mg
  Interventions: Drug: HKI-357
- 5 (Placebo Comparator): 160mg
  Interventions: Drug: HKI-357
- 6 (Placebo Comparator): 240mg
  Interventions: Drug: HKI-357
- 7 (Placebo Comparator): 400mg
  Interventions: Drug: HKI-357
- 8 (Placebo Comparator): 640mg
  Interventions: Drug: HKI-357
- 9 (Placebo Comparator): 960mg
  Interventions: Drug: HKI-357
- 10 (Placebo Comparator): placebo
  Interventions: Drug: HKI-357

INTERVENTIONS:
Drug: HKI-357 — Single-dose capsule

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of single doses of HKI-357 administered to healthy subjects.

ELIGIBILITY:
Eligibility Criteria:

* Healthy adult men or women of nonchildbearing potential, aged 18-50.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, PK | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer